CLINICAL TRIAL: NCT01041859
Title: A Randomized-Withdrawal, Placebo-Controlled, Study Evaluating the Efficacy, Safety, and Tolerability of Tapentadol Extended-Release (ER) in Subjects With Chronic, Painful Diabetic Peripheral Neuropathy (DPN)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Tapentadol ER Compared With Placebo in Patients With Chronic, Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016051; R331333PAI3027 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); KF56 (Other: Grunenthal GmbH)
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-08

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Painful; Polyneuropathy; Peripheral neuropathy
MeSH Terms: conditions — Pain; Polyneuropathies; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol Extended Release (ER) (Experimental)
  Interventions: Drug: Tapentadol extended release (ER)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol extended release (ER) — Type= range, unit= mg, number= 100 to 250, form= tablet, route= oral use. Tapentadol ER optimal dose ranging between 100 mg and 250 mg twice daily for 15 weeks.
  Arms: Tapentadol Extended Release (ER)
Drug: Placebo — Form= tablet, route= oral use. Matching placebo twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of orally administered tapentadol extended release (ER) at dosages of 100 to 250 mg twice daily compared with placebo in patients with moderate to severe pain due to chronic, painful diabetic peripheral neuropathy (DPN) who tolerated tapentadol (ER) and have an initial treatment effect (pain improvement) after a 3-week, open-label titration period.

DETAILED DESCRIPTION:
This is a randomized-withdrawal (only patients that have an initial response to tapentadol are assigned to either tapentadol or placebo), placebo-controlled, multicenter study evaluating the efficacy, safety, and tolerability of orally administered tapentadol, using the extended release tamper-resistant formulation (TRF), at dosages of 100 to 250 mg twice daily in patients with moderate to severe pain due to chronic, painful DPN. The study consists of 1) an open-label (all people involved know the identity of the intervention) phase, including a 13-day screening period, a 5-day washout period (where patients are to stop taking their pain medication), a 3-day pre-titration pain-intensity evaluation period (where patients will record their pain intensity twice daily in the morning and evening), and a 3-week, open-label titration period (all patients receive tapentadol study drug), 2) a 12-week, double-blind (neither physician nor patient knows the name of the assigned drug) maintenance phase, and 3) a posttreatment phase of approximately 10 to 14 days. The study will evaluate the effectiveness of orally administered tapentadol ER versus placebo in reducing patients' pain intensity. The pain intensity will be assessed by comparing the baseline pain level to the level at week 12 of the maintenance phase. The total duration of study drug treatment for each patient will be approximately 15 weeks. Safety and tolerability will be evaluated by vital signs, physical examinations, clinical laboratory tests, 12-lead electrocardiograms (ECGs), standardized neurologic examinations, and monitoring of adverse events. Patients will be titrated on tapentadol ER from a starting dose of 50 mg twice daily to the patient's optimal dose ranging between 100 mg and 250 mg twice a day, or placebo. All doses of study medication will be taken orally with approximately 120 ml of water with or without food for a maximum timeframe of 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or 2 diabetes mellitus must have a documented clinical diagnosis of painful diabetic peripheral neuropathy with symptoms and signs for at least 6 months, and pain present at the time of screening
* Diagnosis must include pain plus reduction or absence of pin sensibility and/or vibration sensibility on Total Neuropathy Score - Nurse (TNSn) examination in lower and/or upper extremities at screening
* The investigator considers the patient's blood glucose to be controlled by diet, or hypoglycemics, or insulin for at least 3 months prior to enrolling in the study
* Patients have been taking analgesic medications for the condition for at least 3 months prior to screening (patients taking opioid analgesics must be dissatisfied with current treatment, and patients taking non-opioid analgesics must be dissatisfied with current analgesia)
* Patients currently requiring opioid treatment must be taking daily doses of an opioid-based analgesic equivalent to <=160mg of oral morphine

Exclusion Criteria:

* Significant history of pulmonary, gastrointestinal, endocrine, metabolic (except diabetes mellitus), neurological, psychiatric disorders (resulting in disorientation, memory impairment or inability to report accurately as in schizophrenia)
* History of moderate to severe hepatic impairment
* Severely impaired renal function
* Clinically significant laboratory abnormalities
* Clinically significant cardiac disease
* History of seizure disorder or epilepsy
* History of any other clinically significant disease that in the investigator's opinion may affect efficacy or safety assessments or may compromise patient safety during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (72):
- United States (60):
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Fresno, California
  - Orange, California
  - Redding, California
  - Sacramento, California
  - San Francisco, California
  - Spring Valley, California
  - Walnut Creek, California
  - Denver, Colorado
  - Clearwater, Florida
  - Hallandale, Florida
  - Miami, Florida
  - Ormond Beach, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Meridian, Idaho
  - Avon, Indiana
  - Evansville, Indiana
  - Fishers, Indiana
  - Prairie Village, Kansas
  - Shreveport, Louisiana
  - Owings Mills, Maryland
  - Pasadena, Maryland
  - Rockville, Maryland
  - Brockton, Massachusetts
  - Edina, Minnesota
  - St Louis, Missouri
  - Cedarhurst, New York
  - Flushing, New York
  - New York, New York
  - Rochester, New York
  - Valley Stream, New York
  - Williamsville, New York
  - Hickory, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Medford, Oregon
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Duncansville, Pennsylvania
  - Anderson, South Carolina
  - Greer, South Carolina
  - Bulverde, Texas
  - Dallas, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Salt Lake City, Utah
  - Alexandria, Virginia
  - Norfolk, Virginia
  - Virginia Beach, Virginia
- Canada (11):
  - Calgary, Alberta
  - Kelowna, British Columbia
  - Barrie, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Hawkesbury, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Dollard-des-Ormeaux, Quebec
  - Laval, Quebec
  - Montreal, Quebec
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In a 3-week open-label (OL) period, patients titrated to an optimal dose between 100 mg and 250 mg twice daily. Patients with >=1-point reduction in pain intensity at the end of OL period were randomized. 38 of 358 who completed OL were not randomized: <1-pt reduction(28), withdrew consent(4), non-compliant(2), adverse events(1), other reason(3).
Groups:
- OL Tapentadol: Tapentadol extended release (ER) 50 100 150 200 250 mg twice daily for 3 weeks
- DB Tapentadol ER: Tapentadol extended release (ER) 100 150 200 250 mg twice daily for 12 weeks
- DB Placebo: Double-Blind Placebo Control Group
Period: Open-Label Titration
Arm/Group | OL Tapentadol | DB Tapentadol ER | DB Placebo
Started | 459 (Of 460 total enrollment, one subject enrolled twice; this subject's second enrollment is excluded.) | 0 | 0
Completed | 358 (Of 358 completed subjects, 320 were randomized to the Double-Blind Maintenance Period.) | 0 | 0
Not Completed | 101 | 0 | 0
Not completed — Adverse Event | 69 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other | 7 | 0 | 0
Not completed — Noncompliance With Study Drug | 8 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0
Period: Double-Blind Maintenance
Arm/Group | OL Tapentadol | DB Tapentadol ER | DB Placebo
Started | 0 | 166 (168 were randomized, 2 were not treated (1 randomized in error, 1 withdrew consent).) | 152 (152 randomized, all were treated.)
Completed | 0 | 120 | 107
Not Completed | 0 | 46 | 45
Not completed — Adverse Event | 0 | 23 | 13
Not completed — Lack of Efficacy | 0 | 3 | 11
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 3
Not completed — Other | 0 | 6 | 2
Not completed — Noncompliance With Study Drug | 0 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Tapentadol ER | DB Placebo | Total
Number analyzed (Participants) | 166 | 152 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 109 | 231
  >=65 years | 44 | 43 | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.63) | 59 (9.00) | 58.7 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 64 | 131
  Male | 99 | 88 | 187
Region Enroll [Number; unit: participants]
  Canada | 24 | 22 | 46
  USA | 142 | 130 | 272

OUTCOME MEASURES:

1. Primary Outcome: Change From Double-Blind Baseline of the Average Pain Intensity Based on an 11-point Numerical Rating Scale(NRS) Over the Last Week of the Maintenance Period at Week 12
Description: For this twice daily pain assessment, the patients were to indicate the level of pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Double-Blind Baseline and 12 weeks (Primary endpoint is the average pain intensity score during the last week of the maintenance period)
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) was used to impute pain score after discontinuation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Tapentadol ER | DB Placebo
Number analyzed (Participants) | 165 | 152
units on a scale | 0.28 (2.04) | 1.3 (2.43)
Statistical Analysis 1: Comparison: DB Tapentadol ER vs DB Placebo; The primary null hypothesis to be tested for the study was that the tapentadol ER group was not different from the placebo group for the primary endpoint. Assuming the mean treatment group difference of 1.0 with an SD of 2.6, 144 subjects per treatment group were estimated to provide 90% power to show that the tapentadol ER group was statistically different from placebo at an alpha level of 0.05. The total number of subjects to be randomly assigned to a DB treatment group for the study was 300; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) model was used with treatment, dose level, and pooled analysis center as factors and baseline pain intensity score as a covariate; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.415 to -0.493], Standard Error of Mean 0.234 — Mean Difference is least squares mean change in DB Tapentadol ER group minus least squares mean change in DB Placebo group (based on ANCOVA model)

2. Secondary Outcome: Responder Analysis: Proportion of Patients With At Least 50% Improvement From Baseline of Open-Label on the Numerical Rating Scale (NRS) at the Week 12 Endpoint
Description: The NRS was a twice-daily pain assessment in which patients were to indicate the level of pain experienced over the previous 12 hours on an 11-point scale with a score of 0 indicating "no pain" and a score of 10 indicating "pain as bad as you can imagine".
Time Frame: Open-label Baseline and End of Double-Blind Treatment at 15 Weeks (3 weeks open-label plus 12 weeks double-blind)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DB Tapentadol ER | DB Placebo
Number analyzed (Participants) | 166 | 152
percentage of participants | 40.4 (2.04) | 28.9 (2.43)

3. Secondary Outcome: Distribution of Patient Global Impression of Change at Week 12 Endpoint
Description: Patient Global Impression of Change (PGIC) is a patient-rated assessment of overall neuropathic pain since the start of treatment using a categorical scale 1-7, where 1 is 'very much improved' and 7 is 'very much worse'
Time Frame: End of Double-Blind Treatment at 12 Weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point
Measure: Number; unit: percentage of participants
Arm/Group | DB Tapentadol ER | DB Placebo
Number analyzed (Participants) | 150 | 139
percentage of participants
  Very much improved | 28.7 (2.04) | 14.4 (2.43)
  Much improved | 37.3 | 30.9
  Minimally improved | 21.3 | 20.9
  Not changed | 8.0 | 18.7
  Minimally worse | 2.0 | 5.0
  Much worse | 1.3 | 7.9
  Very much worse | 1.3 | 2.2

4. Secondary Outcome: Change From Baseline of Open-Label in the Pain Intensity Subscale of the Brief Pain Inventory (BPI) at the Week 12 Double-Blind Endpoint
Description: The BPI is a 12-item questionnaire to evaluate the intensity of pain and the degree to which pain interferes with function. It includes 4 items assessing current pain intensity and pain at its worst, least, and on average over the past day using an 11-point scale from 0 = no pain to 10 = pain as bad as you can imagine. The pain intensity subscale score is defined as the mean of the scores from these 4 items.
Time Frame: Open-label Baseline and End of Double-Blind Treatment at 15 Weeks (3 weeks open-label plus 12 weeks double-blind)
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Tapentadol ER | DB Placebo
Number analyzed (Participants) | 147 | 137
units on a scale | -3.0 (2.16) | -2.3 (2.33)

5. Secondary Outcome: Change From Baseline in the EuroQoL-5 Dimension (EQ-5D) Health Status Index at the Week 12 Endpoint
Description: EQ-5D has 5 items (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) rated on a categorical scale of 1-3 with 1=no problems, 2=some problems, 3=extreme problems. The health state index is a weighted combination of the 5 items. It has a range of 0 to 1, with 0=deceased and 1=full health.
Time Frame: Double-blind Baseline and End of Double-Blind Treatment at 12 Weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Tapentadol ER | DB Placebo
Number analyzed (Participants) | 146 | 135
units on a scale | 0.00 (0.203) | -0.10 (0.257)

ADVERSE EVENTS:
Arm/Group | OL Tapentadol | DB Tapentadol ER | DB Placebo
Serious Adverse Events (participants affected / at risk) | 11/459 | 8/166 | 9/152
Other Adverse Events (participants affected / at risk) | 296/459 | 86/166 | 37/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Tapentadol (N=459) | DB Tapentadol ER (N=166) | DB Placebo (N=152)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic Foot Infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 0
Arterial Stenosis Limb (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 2
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry Gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 3 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram Change (Investigations) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1
Coronary Artery Bypass (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL Tapentadol (N=459) | DB Tapentadol ER (N=166) | DB Placebo (N=152)
Nausea (Gastrointestinal disorders) | 112 | 34 | 14
Vomiting (Gastrointestinal disorders) | 46 | 20 | 6
Diarrhoea (Gastrointestinal disorders) | 24 | 11 | 10
Constipation (Gastrointestinal disorders) | 54 | 9 | 0
Dry Mouth (Gastrointestinal disorders) | 40 | 8 | 2
Dizziness (Nervous system disorders) | 78 | 12 | 2
Somnolence (Nervous system disorders) | 49 | 10 | 1
Headache (Nervous system disorders) | 44 | 4 | 8
Insomnia (Psychiatric disorders) | 14 | 9 | 4
Anxiety (Psychiatric disorders) | 9 | 7 | 8
Fatigue (General disorders) | 44 | 12 | 1
Nasopharyngitis (Infections and infestations) | 5 | 9 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.